CLINICAL TRIAL: NCT03188471
Title: Preventive Application of GnRH Antagonist on Early Ovarian Hyperstimulation Syndrome in High-risk Women: A Prospective Randomized Trial
Brief Title: Preventive Application of GnRH Antagonist on Early OHSS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhou Canquan, Chief of the Center for Reproductive Medicine and Department of Gynecology & Obstetrics, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: antagonist
Record Dates: First submitted 2017-06-10; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Ovarian Hyperstimulation Syndrome; GnRH Antagonist; Aspirin; Vascular Endothelial Growth Factor; Pigment Epithelium Derived Factor
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Aspirin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GnRH antagonist (Experimental): Vitamin C (1 tablet daily) as placebo of aspirin GnRH antagonist 0.25mg daily from the day of oocyte retrieval for seven days
  Interventions: Drug: GnRH antagonist
- aspirin (Active Comparator): aspirin (100 mg daily, plus saline as placebo of GnRH antagonist ) for seven days.
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: GnRH antagonist — GnRH antagonist 0.25mg daily from the day of oocyte retrieval for seven days for high risk of ovarian hyper stimulation syndrome patients
  Other Names: Vitamin C platelet
  Arms: GnRH antagonist
Drug: aspirin — aspirin (100 mg daily, plus saline as placebo of GnRH antagonist ) for seven days
  Other Names: saline as placebo of GnRH antagonist
  Arms: aspirin

SUMMARY:
Ovarian hyperstimulation syndrome is an iatrogenic complication of controlled ovarian stimulation. Ovarian hyperstimulation syndrome prevention is a multistage process and more important than treatment.Preventive administration of GnRH antagonist for high risk OHSS patients from the day of oocyte retrieval is not investigated. Besides, the relevant mechanism is not clear yet. Here we designed a prospective randomized study to investigate whether GnRH anatagonist treatment after oocyte retrieval is more effective in preventing early ovarian hyperstimulation syndrome development than traditional aspirin preventive administration in women at high risk for OHSS.

DETAILED DESCRIPTION:
Ovarian hyperstimulation syndrome is an iatrogenic complication of controlled ovarian stimulation. Early ovarian hyperstimulation syndrome (OHSS) occurs during luteal phase of controlled ovarian stimulation within 9 days after human chorionic gonadotropin trigger and reflects an acute consequence of this hormone on the ovaries.Ovarian hyperstimulation syndrome prevention is a multistage process and more important than treatment.Recently the administration of GnRH antagonists during the luteal phase of in vitro fertilization cycles offers another therapeutic modality for patients with severe early OHSS.However, preventive administration of GnRH antagonist for high risk OHSS patients from the day of oocyte retrieval is not investigated. Besides, the relevant mechanism is not clear yet. Here we designed a prospective randomized study to investigate whether GnRH anatagonist treatment after oocyte retrieval is more effective in preventing early ovarian hyperstimulation syndrome development than traditional aspirin preventive administration in women at high risk for OHSS.

ELIGIBILITY:
Inclusion Criteria:

* number of oocyte retrieval more than 25;
* estradiol level higher than 5000pg/mL on the day of human chorionic gonadotropin administration;
* clinical or ultrasonography proven ovarian hyperstimulation syndrome on the day of oocyte retrieval.

Exclusion Criteria:

* contraindications to GnRH antagonist;
* coasting or other preventive measures for managing ovarian hyperstimulation syndrome had been applied;
* GnRH agonist for trigger.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 175 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of early ovarian hyperstimulation syndrome | up to 1 month
  Incidence and severity of early ovarian hyperstimulation syndrome according to its classification

SECONDARY OUTCOMES:
vascular endothelial growth factor level | up to 1 month
  VEGF level
pigment epithelium derived factor level | up to 1 month
  PEDF level
incidence of hydrothorax | up to 1 month
  one criterion for evaluation of OHSS severity
incidence of liver dysfunction | up to 1 month
  one criterion for evaluation of OHSS severity
incidence of renal dysfunction | up to 1 month
  one criterion for evaluation of OHSS severity
incidence of electrolytic imbalance | up to 1 month
  one criterion for evaluation of OHSS severity
incidence of hemoconcentration | up to 1 month
  one criterion for evaluation of OHSS severity
incidence of elevated WBC | up to 1 month
  one criterion for evaluation of OHSS severity

CONTACTS AND LOCATIONS:
Overall Officials: Qingyun Mai, Principal Investigator — Center for Reproductive Medicine and Department of Gynecology & Obstetrics, First Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital of Sun Yatsen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No